CLINICAL TRIAL: NCT03063346
Title: The Effect of a Protein Hydrolysate on Muscle Strength Recovery in Athletes
Brief Title: The Effect of a Protein Hydrolysate on Muscle Strength Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-001
Record Dates: First submitted 2017-02-02; First posted 2017-02-24 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Muscle Strength Recovery
MeSH Terms: interventions — Protein Hydrolysates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein hydrolysate high dose (Experimental)
  Interventions: Dietary Supplement: Protein hydrolysate high dose
- Protein hydrolysate low dose (Experimental)
  Interventions: Dietary Supplement: Protein hydrolysate low dose
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protein hydrolysate high dose
  Arms: Protein hydrolysate high dose
Dietary Supplement: Protein hydrolysate low dose
  Arms: Protein hydrolysate low dose
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Overtraining is a real problem for (semi-)professional athletes. Overtraining is often caused by the bodies' lack of ability to recover between training. In addition, during high intensity training reactive oxygen species are formed up to 20 fold compared to resting values. This causes increased muscle tissue damage after intense exercise, which slows down recovery. Improving recovery may increase an athlete's ability to reach higher training volumes resulting in establishing a higher performance plateau.

It is known that hydrolyzed proteins have a positive effect on muscle protein synthesis due to its faster absorption rate. Therefore, it is hypothesized that a known protein hydrolysate may have positive effects on strength recovery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (based on their medical history provided during a general health questionnaire)
* Participants are amateur or (semi-) professional athletes in resistance or interval sports (engage in >6 hours of intense physical activity per week).
* Age 18 - 35
* Experience in resistance training

Exclusion Criteria:

* Use of creatine supplements and/or anabolic steroids.
* Allergy to test product/protein
* Allergy to specific protein hydrolysate
* BMI lower than 18 or higher than 30.
* Lack of technique in correctly performing a barbell squat (judged by sports physiologist).
* Recent muscle injury in legs or back less than one month before the start of the study.
* Cardiovascular complications
* Use of medication
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study.
* Abuse of products; alcohol (> 20 alcoholic units per week) and drugs

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Muscle strength recovery | 4 weeks
  difference in peak force between the exhaustion challenge and the recovery challenge, measured with a linear encoder during a squat exercise

SECONDARY OUTCOMES:
Blood lactate buildup | 4 weeks
  in mmol/L, measured trough a finger prick after exhaustion and recovery challenge
Body composition | 4 weeks
  fat percentage, based on 4-point skin fold measurement
Exercise volume | 4 weeks
  amount of repetitions x time taken x power, measured with a linear encoder during squat exercise
Peak force output | 4 weeks
  measured with a linear encoder during the squat exercise

IPD SHARING:
Plan to Share IPD: Undecided